CLINICAL TRIAL: NCT01800799
Title: Use of Urinary Nerve Growth Factor as A Biomarker to Determine Complete Resolution of Bladder Inflammation After Acute Bacterial Cystitis in Women
Brief Title: Urinary NGF as A Biomarker for Acute Bacterial Cystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Director of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCGHUROL007
Record Dates: First submitted 2013-02-19; First posted 2013-02-28 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Urinary Tract Infection
Keywords: Urinary tract infection; Urothelium; Inflammation; Apoptosis
MeSH Terms: conditions — Urinary Tract Infections; Inflammation | interventions — Anti-Infective Agents; Celecoxib; Anti-Inflammatory Agents

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No

ARMS (3):
- UTI (WBC>10 per high power field) (Experimental): 1. Antimicrobial agent (Baktar 800mg h.s.)
  2. Anti-inflammatory agent (Celecoxib 200mg QD)
  Interventions: Drug: Baktar 800mg h.s.; Drug: Celecoxib 200mg QD
- Recurrent UTI (Experimental): 1. Antimicrobial agent (Baktar 800mg h.s.)
  2. Anti-inflammatory agent (Celecoxib 200mg QD)
  Interventions: Drug: Baktar 800mg h.s.; Drug: Celecoxib 200mg QD
- Normal control (No Intervention): Normal control

INTERVENTIONS:
Drug: Baktar 800mg h.s. — Antimicrobial agent (Baktar 800mg h.s.)
  Other Names: Antimicrobial agent
  Arms: Recurrent UTI; UTI (WBC>10 per high power field)
Drug: Celecoxib 200mg QD — Anti-inflammatory agent (Celecoxib 200mg QD)
  Other Names: Anti-inflammatory agent
  Arms: Recurrent UTI; UTI (WBC>10 per high power field)

SUMMARY:
This study will enroll 30 female patients with the first time urinary tract infection (UTI), 30 female patients with recurrent UTI and 10 female without any prior history of UTI or urinary tract pathology will be invited to serve as the controls. Urine samples will be collected in the patients at baseline, 7 days after antibiotics treatment, and 2 weeks, 4 weeks, 8 weeks, and 12 weeks. Urinalysis will be performed at each visit and urine culture will be performed at baseline and at the 2 weeks and 3 months visits. Urine samples at baseline and 3 months will be collected from the controls for comparison.

DETAILED DESCRIPTION:
Recurrent UTI is a very bothersome and a popular problem in the urogynecology clinical practice. According to the International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction, recurrent UTI is defined as at least three symptomatic and medically diagnosed UTI in the previous 12 months. The previous UTI(s) should have resolved prior to a further UTI being diagnosed. Recurrent UTI is one of the most common diagnoses for female pelvic floor dysfunction.

Patients with recurrent UTI might also have bladder irritative symptoms. Previous studies have revealed that patients with recurrent UTI have elevated urinary NGF, suggesting chronic inflammation is present in the bladder of these patients after resolution of UTI. The investigators preliminary results showed that chronic inflammation, urothelial cell apoptosis and impairment of barrier function of urothelial cells could be the underlying pathophysiology of recurrent UTI in women. Chronic inflammation might reside in the bladder wall after resolution of UTI, which might also cause urothelial dysfunction and defective barrier function and UTI will be easy to recur in these patients. This evidence provides a new focus for clinical management and future research of recurrent urinary tract infection.

Based on these knowledge, the investigators hypothesized that chronic inflammation might reside in the bladder wall, which might also cause urothelial dysfunction and defective barrier function. UTI might be easy to recur in these patients with residual chronic bladder inflammation. If the investigators can determine complete resolution of the chronic inflammation after acute cystitis episode, it is possible to inhibit recurrent cystitis through treating the inflammation with anti-inflammatory agents.

Nerve growth factor (NGF) is a small secreted protein which induces the differentiation and survival of particular target neurons. NGF has been implicated as a chemical mediator of pathology-induced changes in C-fiber afferent nerve excitability and reflex bladder activity. The levels of neurotrophic factors including NGF increase in the bladder after spinal cord injury (SCI) and increased levels of NGF have been detected in the lumbosacral spinal cord and dorsal root ganglion of rats after SCI. Chronic administration of NGF into the bladder of rats induces bladder hyperactivity and increases the firing frequency of dissociated bladder afferent neurons. Increased levels of urinary NGF have also been detected in BOO patients exhibiting overactive bladder (OAB) symptoms. Increased bladder tissue NGF was noted in patients with interstitial cystitis/painful bladder syndrome (IC/PBS). Recent research has focused on the urinary NGF levels in detecting OAB and IC/PBS in lower urinary tract dysfunction (LUTD). Evidences have shown that urinary proteins such as NGF and prostaglandin E2 levels increase in patients with OAB, sensory urgency and detrusor overactivity (DO). Patients with OAB-dry and OAB-wet have significantly higher urinary NGF levels compared to the control group and patients with increased bladder sensation. The urinary NGF levels increase physiologically with small scale in the normal subjects at urge to void but increase pathologically with large scale in OAB patients at small bladder volume and at urgency sensation. The urinary NGF levels decrease after antimuscarinic therapy and further decrease after detrusor botulinum toxin injections in refractory OAB. Put together, the urinary NGF levels seem to be a potential biomarker for diagnosis of OAB and the underlying chronic inflammation.

Several urological diseases including bacterial cystitis, lower ureteral stone and urothelial cell carcinoma may develop storage symptoms mimicking OAB or IC/PBS. The urinary NGF levels are also elevated in these disorders. In the previous study the investigators found that UTI may increase NGF production in urine associated with urinary tract stones. Patients with resolution of UTI but also with persistent OAB may have high urinary NGF levels. These results provide evidence that urinary NGF is a product of inflammation in the urinary tract. Therefore, urinary NGF may be considered as a second-line product following urothelial damage or changes of urothelial environment that initiate the sensory nerve excitation and cause bladder hypersensitivity or DO. Measuring urinary NGF is a non-invasive tool to assess chronic inflammatory status and for longitudinal comparison of the treatment.

It is essential to know whether the urinary NGF levels can also increase at acute cystitis episode and the production has a relation with the associated storage symptoms in different stage after antibiotics treatment. This study is designed to measure the urinary NGF levels in patients with acute cystitis and different stages after antibiotics treatment. If the urinary NGF levels have association with the underlying inflammation in the bladder wall, the investigators might use it as a biomarker to determine the status of resolution of the inflammation and provide physicians to decide how long should the investigators treat patients with acute cystitis.

Materials and Methods

This study will enroll 30 female patients with the first time UTI and 30 female patients with recurrent UTI (at least two previous UTI episodes in the latest 12 months) but have a recent acute episode. Ten age-matched women (30 to 50 years old) without any prior history of UTI or urinary tract pathology will be invited to serve as the controls. Urine samples will be collected in the patients at baseline, 7 days after antibiotics treatment, and 2 weeks, 4 weeks, 8 weeks, and 12 weeks after the UTI episode. Urinalysis will be performed at each visit and urine culture will be performed at baseline and at the 2 weeks and 3 months visits. Urine samples at baseline and 3 months will be collected from the controls for comparison.

All patients should be proven to have UTI by detecting pyuria in urinalysis (WBC>10 per high power field) and had a positive urine culture result. In addition, a kidney, ureter, and bladder (KUB) film, and renal sonography will be performed to exclude to possibility of urolithiasis or other urinary tract pathology. The one-day voiding diary will be requested to record at each visit to determine the functional bladder capacity (FBC) and frequency episodes per day. Bladder symptoms will be recorded by Overactive Bladder Symptom Score (OABSS) and visual analog scale of pain (VAS). In addition, uroflowmetry, including maximum flow rate (Qmax), voided volume and postvoid residual volume (PVR) will also be measured at visit 2. Urine samples at baseline and each visit after treatment will be collected at a comfortably full bladder and sent for NGF measurements. Antibiotics (Cephalexin 500mg Q6H) for 1 to 2 weeks will be started at the baseline until the urinalysis proven negative and urine culture turned to be negative. Then antimicrobial agent (Baktar 800mg h.s.) or anti-inflammatory agent (Celecoxib 200mg QD) will be randomly prescribed for UTI prophylaxis for 3 months after complete resolution of acute cystitis. All patients will be followed-up for up to one year to monitor whether they have occurrence of recurrent UTI.

All urine samples will be collected with a full bladder and natural voiding. Measurement of urinary NGF levels will be performed by the ELISA method. Urine samples are not diluted. Voided urine is put on ice immediately and centrifuged at 3000 g for 10 min at 4 ◦C. The supernatant is separated into aliquots in 1.5 mL tubes and preserved in a -80 ◦C freezer. At the same time, 3 mL of urine is taken to measure urinary creatinine levels. Urinary NGF concentration is determined using the Emax ImmunoAssay System (Promega, Madison, Wisconsin, USA) with a specific and highly sensitive ELISA kit, which has a minimum sensitivity of 7.8 pg/mL. The amount of NGF in urine samples fall below the detection limits of NGF assay was extracted from an NGF standard curve. All samples will be run in triplicate, urinary NGF levels without a consistent value in three measures will be repeated and the values will be averaged. The total urinary NGF levels are further normalized by the concentration of urinary creatinine (NGF/Cr level). The NGF/Cr levels are compared among all subgroups.

Statistical analyses will be performed by a paired t-test for paired data in consecutive time points. Mann-Whitney test will be used for non-parametric analysis between different subgroups. A P-value of less than 0.05 is considered significant.

Expected Results

The investigators hypothesized that patients with recurrent UTI may have persistently elevated urinary NGF levels compared with those with the first time UTI. The urinary NGF levels will remain elevated in patients who have persistent OAB symptoms after acute cystitis episode and might be persistently higher than the controls after 3 months. Patients treated with anti-inflammatory agent might have lower urinary NGF levels at 3 months visit compared to those taking antimicrobials. The incidence of recurrent UTI in the following one year might be more in the patients treating with antimicrobials than those treating with anti-inflammatory agents.

ELIGIBILITY:
Inclusion Criteria:

* Female adults aged ≥ 20 years.
* All patients should be proven to have UTI by detecting pyuria in urinalysis (WBC>10 per high power field) and had a positive urine culture result.
* A KUB film, and renal sonography will be performed to exclude to possibility of urolithiasis or other urinary tract pathology.
* Not yet have lower urinary tract surgery in the past.
* The patient has not yet accepted anticholinergic medication
* Patient or his legally acceptable representative has signed the written informed consent form.

Exclusion Criteria:

* Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up.
* Patients with uncontrolled confirmed diagnosis of acute urinary tract infection.
* Patients have laboratory abnormalities at screening including: (1) Aspartate aminotransferase (AST) > 3 x upper limit of normal range. (2) Alanine aminotransferase (ALT) > 3 x upper limit of normal range. (3) Patients have abnormal serum creatinine level > 2 x upper limit of normal range.
* Female patients who is pregnant, lactating, or with child-bearing potential without contraception.
* Patients with any other serious disease or condition considered by the investigator not suitable for entry into the trial.
* Patients participated investigational drug trial within 1 month before entering this study.
* Patient or his legally written informed consent hadn't been obtained.

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in urinary nerve growth factor (NGF) at different time points | 1 week, 1 month, 2 months and 3 months
  Change from Baseline in urinary nerve growth factor (NGF) at different time points (1 week, 1 month, 2 months and 3 months).

SECONDARY OUTCOMES:
Change from Baseline in one-day voiding diary at different time points | 1 week, 1 month, 2 months and 3 months
  Change from Baseline in one-day voiding diary at different time points (1 week, 1 month, 2 months and 3 months).
  The one-day voiding diary will be requested to record at each visit to determine the functional bladder capacity (FBC) and frequency episodes per day.
Change from Baseline in Overactive Bladder Symptom Score (OABSS) at different time points | 1 week, 1 month, 2 months and 3 months
  Change from Baseline in Overactive Bladder Symptom Score (OABSS) at different time points (1 week, 1 month, 2 months and 3 months).
Change from Baseline in visual analog scale of pain (VAS) at different time points | 1 week, 1 month, 2 months and 3 months
  Change from Baseline in visual analog scale of pain (VAS) at different time points (1 week, 1 month, 2 months and 3 months).

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital and Tzu Chi University
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Liu HT, Chen CY, Kuo HC. Urinary nerve growth factor levels in overactive bladder syndrome and lower urinary tract disorders. J Formos Med Assoc. 2010 Dec;109(12):862-78. doi: 10.1016/S0929-6646(10)60133-7. PMID 21195884
- [Background] Vizzard MA. Changes in urinary bladder neurotrophic factor mRNA and NGF protein following urinary bladder dysfunction. Exp Neurol. 2000 Jan;161(1):273-84. doi: 10.1006/exnr.1999.7254. PMID 10683293
- [Background] Yoshimura N. Bladder afferent pathway and spinal cord injury: possible mechanisms inducing hyperreflexia of the urinary bladder. Prog Neurobiol. 1999 Apr;57(6):583-606. doi: 10.1016/s0301-0082(98)00070-7. PMID 10221783
- [Background] Vizzard MA. Neurochemical plasticity and the role of neurotrophic factors in bladder reflex pathways after spinal cord injury. Prog Brain Res. 2006;152:97-115. doi: 10.1016/S0079-6123(05)52007-7. PMID 16198696
- [Background] Seki S, Sasaki K, Igawa Y et al. Detrusor overactivity induced by increased levels of nerve growth factor in bladder afferent pathways in rats. Neurourol Urodyn 2003; 22: 375-7
- [Background] Lamb K, Gebhart GF, Bielefeldt K. Increased nerve growth factor expression triggers bladder overactivity. J Pain. 2004 Apr;5(3):150-6. doi: 10.1016/j.jpain.2004.01.001. PMID 15106127
- [Background] Yoshimura N, Bennett NE, Hayashi Y, Ogawa T, Nishizawa O, Chancellor MB, de Groat WC, Seki S. Bladder overactivity and hyperexcitability of bladder afferent neurons after intrathecal delivery of nerve growth factor in rats. J Neurosci. 2006 Oct 18;26(42):10847-55. doi: 10.1523/JNEUROSCI.3023-06.2006. PMID 17050722
- [Background] Zvara P, Vizzard MA. Exogenous overexpression of nerve growth factor in the urinary bladder produces bladder overactivity and altered micturition circuitry in the lumbosacral spinal cord. BMC Physiol. 2007 Aug 28;7:9. doi: 10.1186/1472-6793-7-9. PMID 17725832
- [Background] Liu HT, Kuo HC. Urinary nerve growth factor levels are increased in patients with bladder outlet obstruction with overactive bladder symptoms and reduced after successful medical treatment. Urology. 2008 Jul;72(1):104-8; discussion 108. doi: 10.1016/j.urology.2008.01.069. Epub 2008 Apr 8. PMID 18400272
- [Background] Lowe EM, Anand P, Terenghi G, Williams-Chestnut RE, Sinicropi DV, Osborne JL. Increased nerve growth factor levels in the urinary bladder of women with idiopathic sensory urgency and interstitial cystitis. Br J Urol. 1997 Apr;79(4):572-7. doi: 10.1046/j.1464-410x.1997.00097.x. PMID 9126085
- [Background] Liu HT, Kuo HC. Intravesical botulinum toxin A injections plus hydrodistension can reduce nerve growth factor production and control bladder pain in interstitial cystitis. Urology. 2007 Sep;70(3):463-8. doi: 10.1016/j.urology.2007.04.038. PMID 17905097
- [Background] Kim JC, Park EY, Seo SI, Park YH, Hwang TK. Nerve growth factor and prostaglandins in the urine of female patients with overactive bladder. J Urol. 2006 May;175(5):1773-6; discussion 1776. doi: 10.1016/S0022-5347(05)00992-4. PMID 16600756
- [Background] Liu HT, Chancellor MB, Kuo HC. Urinary nerve growth factor levels are elevated in patients with detrusor overactivity and decreased in responders to detrusor botulinum toxin-A injection. Eur Urol. 2009 Oct;56(4):700-6. doi: 10.1016/j.eururo.2008.04.037. Epub 2008 Apr 30. PMID 18472208
- [Background] Liu HT, Kuo HC. Urinary nerve growth factor level could be a potential biomarker for diagnosis of overactive bladder. J Urol. 2008 Jun;179(6):2270-4. doi: 10.1016/j.juro.2008.01.146. Epub 2008 Apr 18. PMID 18423678
- [Background] Liu HT, Kuo HC. Urinary nerve growth factor levels are elevated in patients with overactive bladder and do not significantly increase with bladder distention. Neurourol Urodyn. 2009;28(1):78-81. doi: 10.1002/nau.20599. PMID 19089891
- [Background] Liu HT, Chancellor MB, Kuo HC. Decrease of urinary nerve growth factor levels after antimuscarinic therapy in patients with overactive bladder. BJU Int. 2009 Jun;103(12):1668-72. doi: 10.1111/j.1464-410X.2009.08380.x. Epub 2009 Feb 11. PMID 19220267
- [Background] Kuo HC, Liu HT, Tyagi P, Chancellor MB. Urinary Nerve Growth Factor Levels in Urinary Tract Diseases With or Without Frequency Urgency Symptoms. Low Urin Tract Symptoms. 2010 Sep;2(2):88-94. doi: 10.1111/j.1757-5672.2010.00065.x. Epub 2010 May 3. PMID 26676289